CLINICAL TRIAL: NCT02490397
Title: Impact of Daylight on Period 2 Protein and Glycolytic Enzymes in Human Buccal Mucosa and Blood Samples
Brief Title: Impact of Daylight on Patients With Acute Myocardial Infarction
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: not enough participants
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-1607
Record Dates: First submitted 2015-06-24; First posted 2015-07-03 (Estimated); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Coronary Arteriosclerosis; Myocardial Infarction
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exposed to Day light (Experimental): Patients with myocardial infarction (MI): This group will be enrolled on the day of their MI. A blood draw will be performed before any light therapy. The patients will then receive a light box (Square One Wake Up Light NatureBright 10,000 LUX) that they shall use every morning from 8.30-9.00 AM for the next 2 weeks. At the conclusion of the two weeks another blood sample will be drawn.
  Interventions: Other: Day Light
- Exposed to Room light (Sham Comparator): Patients with myocardial infarction (MI): This group will be enrolled on the day of their MI and will only be exposed to room light. They will have blood drawn on the day of enrollment and then at 2 weeks after the MI.
  Interventions: Other: Room Light

INTERVENTIONS:
Other: Day Light — Patients are exposed to day light for 2 weeks after a heart attack. At the end of 2 weeks they will have blood drawn.
  Other Names: Active
  Arms: Exposed to Day light
Other: Room Light — Patients will be exposed to only room or natural light for 2 weeks after heart attack. At the end of 2 weeks they will have blood drawn.
  Other Names: Control
  Arms: Exposed to Room light

SUMMARY:
The study tests if intense light could be a potential therapy in humans after myocardial infarction by inducing Per2.

DETAILED DESCRIPTION:
Damage to the heart caused by a myocardial infarction (heart attack) occurs most often during the early morning hours (6AM). Thus, the involvement of the circadian system (circa= approximately day) has been suggested. The circadian system in humans or animals is based on the rotation of the earth with day and night phases. When humans (or animals) wake up light shines in their eyes and the body receives a signal that the day starts. For the human body it means that certain proteins (named clock, period etc) are produced. The protein that determines the length of a day (awake and sleep period) is called Period 2 (Per2). Recent data indicated that the Per2 protein in hearts from mice is induced after daylight exposure (daylight with an intensity comparable to a bright day at the beach was used, approx. 10 000 LUX). This more Per2 was able to protect the heart from being damaged by no blood going to the heart (protection from a heart attack). This protection was based on a more efficient use of sugars (carbohydrates). Thereby the heart needs less oxygen. Current data indicate that human Per2 is also induced by light exposure and can be detected in human plasma samples.

In this study Per2 transcript and protein levels will be analyzed in patients that just experienced a heart attack with and without intense light (daylight) therapy utilizing blood samples (erythrocytes and leukocytes).

ELIGIBILITY:
Inclusion Criteria:

* Patients with an acute myocardial infarction
* Healthy volunteers
* Must speak and understand English

Exclusion Criteria:

* Patients with an acute myocardial infarction but are too sick, e.g. severe symptoms, chest pain, generally unstable, etc.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-07; Primary Completion 2020-12-28 (Actual); Study Completion 2020-12-28 (Actual)

PRIMARY OUTCOMES:
Change of Period 2 (Per2) protein levels | 2 weeks
  Measure of Per2 protein levels related to daylight exposure vs. room light exposure after 2 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Eckel, MD, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver | Anschutz Medical Campus, Denver, Colorado, United States

REFERENCES:
- [Background] Brainard J, Gobel M, Scott B, Koeppen M, Eckle T. Health implications of disrupted circadian rhythms and the potential for daylight as therapy. Anesthesiology. 2015 May;122(5):1170-5. doi: 10.1097/ALN.0000000000000596. No abstract available. PMID 25635592
- [Background] Brainard J, Gobel M, Bartels K, Scott B, Koeppen M, Eckle T. Circadian rhythms in anesthesia and critical care medicine: potential importance of circadian disruptions. Semin Cardiothorac Vasc Anesth. 2015 Mar;19(1):49-60. doi: 10.1177/1089253214553066. Epub 2014 Oct 7. PMID 25294583
- [Background] Eckle T, Hartmann K, Bonney S, Reithel S, Mittelbronn M, Walker LA, Lowes BD, Han J, Borchers CH, Buttrick PM, Kominsky DJ, Colgan SP, Eltzschig HK. Adora2b-elicited Per2 stabilization promotes a HIF-dependent metabolic switch crucial for myocardial adaptation to ischemia. Nat Med. 2012 Apr 15;18(5):774-82. doi: 10.1038/nm.2728. PMID 22504483